CLINICAL TRIAL: NCT00388570
Title: A Multicenter, Device Randomized, Open-label Prospective Single-cohort Study of Monitoring Exhaled NO in Symptomatic Asthmatic Adults and Children During Anti-inflammatory Treatment
Brief Title: Study of Monitoring Exhaled NO in Symptomatic Asthmatic Adults and Children During Anti-inflammatory Treatment
Acronym: eNOugh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerocrine AB (Industry)
Responsible Party: Aerocrine AB, Ulrika Stein Grive, Aerocrine AB
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: AER-036
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: Asthma; adult; paediatric; NIOX MINO®; NIOX®; nitric oxide; airway inflammation; open-label; single-cohort
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Aerocrine NIOX MINO® Airway Inflammation Monitor

SUMMARY:
The purpose of this study is to demonstrate substantial equivalence between two medical devices which measure nitric oxide in exhaled breath, NIOX MINO® and NIOX® in Symptomatic Asthmatic Adults and Children.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways. Chronically inflamed airways are hyperresponsive; they become obstructed and airflow is limited (by bronchoconstriction, mucus plugs, and increased inflammation) when airways are exposed to various risk factors. Asthma causes recurring episodes of wheezing, breathlessness, chest tightness, and coughing particularly at night or in the early morning.

NO is an important endogenous regulatory molecule that is widely distributed throughout the body. The detection of NO in exhaled air was first reported in 1991, and, soon after it was shown that the levels NO in exhaled air are elevated in patients with asthma. There is now much evidence showing that measurement of the concentration of NO in exhaled air offers a useful non-invasive method of assessing inflammatory airway disease.

Exhaled NO is not increased during bronchospasm unless there is coexisting inflammation. Exhaled NO may have a valuable role in differentiating between the inflammatory and bronchospastic components of clinical asthma, and is also useful for guiding the therapeutic use of steroids and other anti-inflammatory agents.

A study on asthmatics and non-asthmatics subjects has shown that substantial equivalence exists between the stationary device NIOX® and the hand held device NIOX MINO® when comparing NO measurements, when similar conditions are considered and examinations are made as consistently as possible.

In a study with the stationary device NIOX®, exhaled NO was measured before and after two weeks of inhaled corticosteroid treatment in unstable steroid-naïve adult and paediatric asthmatic subjects. The result was a 50.5% mean reduction of exhaled NO. The change in exhaled NO was also compared to change in standard asthma outcome measures, asthma symptoms and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Children, and adults.
* A history of physician-diagnosed asthma or asthma diagnosed by a physician.
* Spirometry performed parameters.
* An increased FENO value.
* Symptomatic asthma as defined on the Asthma Control Questionnaire® (ACQ).

Exclusion Criteria:

* Use of oral corticosteroids.
* Use of intranasal corticosteroids.
* Use of non-steroidal anti-asthma drugs.
* Current serious conditions and/or therapies that are confounding factors.
* Pregnancy.
* Other significant respiratory diseases and/or cardiovascular diseases.
* Current participation in another interventional clinical study.
* Inability to comply with the study procedures, e.g. spirometry and FENO measurements according to standard procedures.
* Unwillingness to sign informed consent and comply with treatment and visits.
* Smoking within 6 months before the study, or a smoking history of >10 pack years or an equivalent amount of other tobacco use.
* Known alcohol or drug abuser.
* Food and beverage (other than water) intake within 1 hour before first FENO measurement
* Nicotine (including nicotine chewing gum, nicotine patch, snuff etc) use within 1 hour before first FENO measurement.
* Strenuous exercise within 1 hour before first FENO measurement

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary analysis variable will be the percent change in FENO measured with
NIOX MINO® and NIOX® between Visit 1 to Visit 2.

SECONDARY OUTCOMES:
Agreement between NIOX MINO® and NIOX® will be assessed by comparing
individual pair-wise FENO measurements from visit V1.
The change in FENO measured with NIOX MINO following corticosteroid therapy
in asthma will be compared with improvements in standard asthma outcome
measures (asthma symptoms and spirometry).
To investigate the inter-operator variability FENO measurements with
NIOX MINO in the same subject when different operators take FENO measurements. Three operator each takes two completed measurements in the same subject in a point of care setting.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Professor, Study Chair — Dept of General Practice and Primary Care, University of Aberdeen; Sven-Erik Dahlén, Professor, Study Chair — Unit for Experimental Asthma and Allergy Research Division of Physiology, The National Institute of Environmental Medicine Karolinska Institutet
Locations (2):
- Näsets Läkargrupp, Falsterbov. 79, SE-23651 Höllviken, Höllviken, Sweden
- Department of General Practice & Primary Care University of Aberdeen, Aberdeen, United Kingdom